CLINICAL TRIAL: NCT04711746
Title: Is Clonal Hematopoiesis of Indeterminate Potential Associated With Unprovoked Pulmonary Embolism?
Acronym: HEMEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PI2020_843_0117
Record Dates: First submitted 2021-01-13; First posted 2021-01-15 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Pulmonary Embolism; Hematopoiesis
Keywords: Pulmonary Embolism; hematopoiesis; genetic sequencing; endothelial dysfunction
MeSH Terms: conditions — Pulmonary Embolism | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Previous proximal unprovoked pulmonary embolism (Experimental)
  Interventions: Biological: blood sample
- Previous proximal provoked pulmonary embolism (Active Comparator)
  Interventions: Biological: blood sample

INTERVENTIONS:
Biological: blood sample — Blood sample withdrawal in order to perform DNA sequencing

SUMMARY:
The clonal hematopoiesis of indetermined prognosis (CHIP) has been described as risk factor for juvenile atherosclerosis. Moreover, some of CHIP genes are responsible of myeloproliferative disorders. Venous thrombosis are frequent in these disorders. The purpose of this project is to determine if CHIP is frequent in unprovoked pulmonary embolism and could be part of the pathophysiology.

ELIGIBILITY:
Inclusion Criteria:

* For cases : Previous proximal unprovoked pulmonary embolism, negative thrombophilia screening.
* For control : Previous proximal provoked pulmonary embolism, negative thrombophilia screening.

Exclusion Criteria:

* Age superior to 65 years old,
* Active cancer

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 544 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Variation of CHIP markers between patients groups | up to 2 years
  Variation of CHIP markers (clonal hematopoiesis of indetermined prognosis ) between patients groups.
  CHIP concept have been defined as a mutation of preleukemic genes at an allelic variation inferior to 2% associated with normal complete blood count.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No